CLINICAL TRIAL: NCT02037620
Title: Recovery of Cardiovascular Function With Epidural Stimulation After Human Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Susan Harkema, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13.0625 CV Epi; ES2-CHN-2013(SH) (Other Grant/Funding Number: CDRF)
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Spinal Cord Injury
Keywords: Epidural Stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Epidural Stimulation (Experimental): 80 sessions each of epidural spinal cord stimulation for 1) cardiovascular function; 2) voluntary movement; and 3) standing.
  Interventions: Device: 5-6-5 Specify electrode; Device: Restore Advance Pulse Generator

INTERVENTIONS:
Device: 5-6-5 Specify electrode
Device: Restore Advance Pulse Generator

SUMMARY:
We propose to demonstrate that epidural stimulation (ES) can be used to recover significant levels of autonomic control of cardiovascular and respiratory function as well as the ability to voluntarily control leg movements below the injury level. This intervention would provide an immediate therapeutic alternative to individuals who now have no recourse for treatment.

DETAILED DESCRIPTION:
We will enroll 4 research participants who have sustained a motor complete SCI to participate in the proposed experiments. Participants will be screened for eligibility, followed by 80 days of usual care, epidural implantation, 80 days of cardiovascular epidural stimulation training, 80 days of voluntary movement (VM) epidural stimulation training and finally 80 days of stand epidural stimulation training. These interventions are done in sequential order, however they are cumulative. In between each intervention, participants will undergo motor and cardiovascular experiments and assessments.

ELIGIBILITY:
1. non-progressive SCI with complete motor paralysis above T1; American Spinal Injury Association Impairment Scale (AIS) A, B or C;
2. 21 - 70 years of age;
3. greater than 2 years post injury;
4. stable medical condition;
5. unable to voluntarily move all single joints of the legs;
6. cardiovascular dysfunction including presence of persistent resting blood pressures and/or symptoms of autonomic dysreflexia and/or orthostatic hypotension; and
7. respiratory dysfunction including at least 15% deficit in predicted pulmonary function outcomes;

Exclusion Criteria:

1. ventilator dependent;
2. painful musculoskeletal dysfunction, unhealed fracture, contracture, or pressure sore that might interfere with training;
3. clinically significant depression or ongoing drug abuse;
4. cardiovascular, respiratory, bladder, or renal disease unrelated to SCI;
5. severe anemia (Hgb<8 g/dl) or hypovelemia; and
6. HIV or AIDS related illness.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Harkema, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Background] Aslan SC, Legg Ditterline BE, Park MC, Angeli CA, Rejc E, Chen Y, Ovechkin AV, Krassioukov A, Harkema SJ. Epidural Spinal Cord Stimulation of Lumbosacral Networks Modulates Arterial Blood Pressure in Individuals With Spinal Cord Injury-Induced Cardiovascular Deficits. Front Physiol. 2018 May 18;9:565. doi: 10.3389/fphys.2018.00565. eCollection 2018. PMID 29867586
- [Background] Mesbah S, Angeli CA, Keynton RS, El-Baz A, Harkema SJ. A novel approach for automatic visualization and activation detection of evoked potentials induced by epidural spinal cord stimulation in individuals with spinal cord injury. PLoS One. 2017 Oct 11;12(10):e0185582. doi: 10.1371/journal.pone.0185582. eCollection 2017. PMID 29020054
- [Result] Harkema SJ, Legg Ditterline B, Wang S, Aslan S, Angeli CA, Ovechkin A, Hirsch GA. Epidural Spinal Cord Stimulation Training and Sustained Recovery of Cardiovascular Function in Individuals With Chronic Cervical Spinal Cord Injury. JAMA Neurol. 2018 Dec 1;75(12):1569-1571. doi: 10.1001/jamaneurol.2018.2617. PMID 30242310
- [Result] Harkema SJ, Wang S, Angeli CA, Chen Y, Boakye M, Ugiliweneza B, Hirsch GA. Normalization of Blood Pressure With Spinal Cord Epidural Stimulation After Severe Spinal Cord Injury. Front Hum Neurosci. 2018 Mar 8;12:83. doi: 10.3389/fnhum.2018.00083. eCollection 2018. PMID 29568266

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidural Stimulation: 80 sessions each of epidural spinal cord stimulation for 1) cardiovascular function; 2) voluntary movement; and 3) standing.
  5-6-5 Specify electrode
  Restore Advance Pulse Generator
Period: Overall Study
Arm/Group | Epidural Stimulation
Started | 5
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Epidural Stimulation
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Blood Pressure in Response to Epidural Stimulation
Description: Noninvasive continuous blood pressure measured from a finger cuff by plethysmographic technique (Finometer Pro, FMS, Amsterdam, Netherlands) was calibrated to brachial blood pressure. Mean arterial pressure was calculated as one-third of systolic blood pressure plus two-third of diastolic blood pressure.
Time Frame: 20 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Epidural Stimulation
Number analyzed (Participants) | 4
mmHg | 112.5 (8.25)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Epidural Stimulation: 80 sessions each of epidural spinal cord stimulation for 1) cardiovascular function; 2) voluntary movement; and 3) standing.
  5-6-5 Specify electrode
  Restore Advance Pulse Generator
  *Each participant received all of the interventions. Thus, adverse events cannot be reported for each independent intervention.
Arm/Group | Epidural Stimulation
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural Stimulation (N=5)
Incision Dehiscence (Surgical and medical procedures) | 3 (3)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epidural Stimulation (N=5)
Right Knee Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/20/NCT02037620/Prot_ICF_000.pdf